CLINICAL TRIAL: NCT01571375
Title: The Differences Between Out-of-hospital Severe Traumatic Brain Injury (TBI) Treatment in a Physician-staffed Versus Paramedic-staffed Emergency Medical Service (EMS) Unit and Its Effect on Patient Prognosis
Brief Title: The Effect of Different Emergency Medical Systems on the Prognosis of Traumatic Brain Injury - a Prospective Study
Status: Suspended | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R10037
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; HEMS; Out-of-hospital; Finland
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FinnHEMS10: Patients Treated by Helsinki HEMS.
- FinnHEMS30: PAtients Treated by Tampere HEMS.

SUMMARY:
The Aim of the Study is to Measure the Effect of Finnish Physician-staffed EMS Unit Treatment Methods on Traumatic Brain Injury (TBI) Patient Prognosis.

Physician-staffed HEMS unit was implemented to the EMS 2011. The aim of this study is to compare the results against a historical database to see if the implementation of a HEMS unit will improve the prognosis of TBI patients.

DETAILED DESCRIPTION:
A Secondary Aim is to Identify Out-of-hospital Treatment Factors That Can be Influenced by Education and Protocols.

ELIGIBILITY:
Inclusion Criteria:

* TBI with CGS < 9 or unconsciousness verified by an on-call neurosurgeon during admission to the hospital.

Exclusion Criteria:

* Multiple trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-06; Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year

SECONDARY OUTCOMES:
Glasgow Outcome Score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, professor, Study Director — Tampere University Hospital; Tom Silfvast, PhD, Study Director — Helsinki University Central Hospital; Tarja Randell, PhD, Study Chair — Helsinki University Central Hospital; Ilkka Virkkunen, PhD, Study Chair — Tampere University Hospital; Toni Pakkanen, M.D., Principal Investigator — Tampere University
Locations (1):
- Tampere University Hospital, Tampere, Finland